CLINICAL TRIAL: NCT04514081
Title: A Randomized, Open-label, Phase 2 Trial of Chidamide+Decitabine+Camrelizumab Versus Decitabine+Camrelizumab in Anti-PD-1 Antibody Resistant Patients With Classical Hodgkin Lymphoma.
Brief Title: The Clinical Trial of Chidamide+Decitabine+Camrelizumab Versus Decitabine+Camrelizumab in Anti-PD-1 Antibody Resistant Patients With Classical Hodgkin Lymphoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-057
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Hodgkin Lymphoma; Anti-PD-1 Antibody Resistant
MeSH Terms: conditions — Hodgkin Disease | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Decitabine; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chidamide+Decitabine+Camrelizumab (Experimental)
  Interventions: Drug: Chidamide; Decitabine; Camrelizumab
- Decitabine+Camrelizumab (Active Comparator)
  Interventions: Drug: Decitabine+Camrelizumab

INTERVENTIONS:
Drug: Chidamide; Decitabine; Camrelizumab — Chidamide is a novel and orally active benzamide class of HDAC inhibitor that selectively inhibits activity of HDAC1, 2, 3 and 10, which can Induce tumor-cell apoptosis, suppress cell proliferation and enhance immune surveillance.
  Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1(DNMT1), which can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function.
  Camrelizumab is a humanized anti-PD-1 monoclonal antibody.
  Arms: Chidamide+Decitabine+Camrelizumab
Drug: Decitabine+Camrelizumab — Decitabine+Camrelizumab
  Arms: Decitabine+Camrelizumab

SUMMARY:
This open-label, randomized, two-arm, phase 2 study has the primary objective of comparing the ORR obtained with Chidamide+Decitabine+Camrelizumab against that obtained with Decitabine+Camrelizumab in patients with Hodgkin Lymphoma who were confirmed resistant to Anti-PD-1 antibody therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological confirmation of relapsed or refractory Hodgkin lymphoma (HL).
2. 12 to 75 years of age.
3. ECOG performance of less than 2.
4. Life expectancy of at least 3 months.
5. Subjects with lymphoma must have at least one measureable lesion >1 cm as defined by lymphoma response criteria.
6. Subjects must have received Anti-PD-1 antibody therapy and were confirmed Anti-PD-1 antibody resistant. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months.
7. Subjects must have adequate marrow, live, renal and heart functions.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in 1 month.
4. Prior organ allograft.
5. Women who are pregnant or breastfeeding.
6. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
7. Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR assess by investigators per the 2014 Lugano classification | 3 years
  rate of subjects achieved objective response in all evaluable subjects
Number of Subjects with treatment-related adverse events (AEs) | 3 years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China